CLINICAL TRIAL: NCT02042599
Title: Pharmacokinetic Study of 48-hour Sevoflurane Inhalation Using a Disposable Delivery System (AnaConDa©) in ICU Patients With Acute Kidney Injury
Acronym: SEVOKID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0175; 2012-005746-37
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Acute Kidney Injury
Keywords: Pharmacokinetics; Sevoflurane; Acute kidney injury; Sedation; ICU patients
MeSH Terms: conditions — Acute Kidney Injury | interventions — Intensive Care Units

ARMS (1):
- sevoflurane (Experimental): Determination of plasmatic concentrations of sevoflurane at different times of a 48h sedation of sevoflurane in ICU patients with acute kidney injury
  Interventions: Drug: Sedation with sevoflurane during 48-hr in ICU

INTERVENTIONS:
Drug: Sedation with sevoflurane during 48-hr in ICU
  Other Names: Determination of plasmatic concentrations of sevoflurane at different times of a 48h sedation of sevoflurane in ICU patients with acute kidney injury

SUMMARY:
Describing a pharmacokinetic model of 48-h sevoflurane sedation in ICU patients with acute kidney failure

DETAILED DESCRIPTION:
Prospective clinical monocentric study in ICU with sedated ventilated patients (presenting acute kidney failure) with sevoflurane during 48 h with the AnaConda® system, establishing pharmacokinetic model of sevoflurane and its metabolites (hydroxyfluroisopropanol, fluoride)

ELIGIBILITY:
Inclusion Criteria:

- Adult patients ventilated more than 48 h Stable respiratory and hemodynamic conditions Consent of patients or family Arterial line AKIN score = 3

Exclusion Criteria:

* BMI <30 Sevoflurane anaphylaxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Determination of plasmatic concentrations of sevoflurane before using AnaConda® system | at 5min, 60 min, 24 hrs and just before the end of sedation.

SECONDARY OUTCOMES:
Determination of plasmatic concentrations of HFIP and fluoride | at 5min, 15 min, 60 min and just before the end of sedation. And 5 min, 10 min, 30 min, 120 min and 360 min after the end of sedation

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France